CLINICAL TRIAL: NCT04469387
Title: Preventive Effect of Limited Decompression on Adjacent Segment With Pre-existing Spinal Canal Stenosis Following Posterior Lumbar Interbody Fusion: a Prospective Interventional Study
Brief Title: Preventive Effect of Limited Decompression on Adjacent Segment Following Posterior Lumbar Interbody Fusion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M2020285
Record Dates: First submitted 2020-07-08; First posted 2020-07-14 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-06

CONDITIONS: Degenerative Lumbar Spinal Stenosis; Degenerative Disc Disease; Degeneration Spine
Keywords: Adjacent segment degeneration; Adjacent segment disease; Pre-existing degeneration; Limited decompression
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NS Group (Active Comparator): NS Group includes patients who simply receive responsible segments fused (L4-S1).
  Interventions: Procedure: Responsible segments fused
- LD Group (Experimental): LD Group includes patients who receive responsible segments fused (L4-S1) plus limited decompression at adjacent segment (L3/4).
  Interventions: Procedure: Limited decompressions at adjacent segment with asymptomatic pre-existing spinal canal stenosis; Procedure: Responsible segments fused

INTERVENTIONS:
Procedure: Limited decompressions at adjacent segment with asymptomatic pre-existing spinal canal stenosis — In terms of limited decompression at the adjacent segment, partial laminotomy, flavectomy, and bilateral medial facetectomies up to the pedicle will be performed. Complete laminectomy and destroy of posterior ligament complex will be avoided.
  Arms: LD Group
Procedure: Responsible segments fused — In terms of responsible segments fused, L4-5 and L5-S1 were fused using posterior lumbar interbody fusion (PLIF).

SUMMARY:
This is a prospective single-center study. Patients requiring posterior lumbar interbody fusion (PLIF) for degenerative disease are prospectively enrolled and followed. Patients enrolled in this study have asymptomatic pre-existing spinal canal stenosis at adjacent segment. This study will focus on the effects of preventative limited decompression at adjacent segment.

DETAILED DESCRIPTION:
Adjacent segment pathologies (ASP), including radiological adjacent segment degeneration (ASDeg) and adjacent segment disease (ASDis) after lumbar fusion surgeries have been troubling complications. The development of ASDis greatly reduces postoperative quality of life, and revision surgery may be required in severe cases. Several risk factors for ASP have been reported, such as age, sex, pre-existing adjacent degeneration, multilevel fusions, sagittal imbalance, the type of fusion, facet tropism and laminar inclination. Previous studies have reported asymptomatic pre-existing spinal canal stenosis (SCS) as a risk factor for ASDis that requires additional surgery. Appropriate strategy needs to be explored for the treatment of asymptomatic pre-existing spinal canal stenosis.

Limited decompressions, including partial laminotomy and flavectomy, have been proved to have the role of enlargement in spinal canal. Therefore, we hypothesize that limited decompressions at adjacent segment with asymptomatic pre-existing SCS will have the preventive effect on ASP.

This prospective study will be limited to patients with the same preoperative pathology, the same fusion segments (L4-5 and L5-S1), the same fusion technique (PLIF). Dynamic X-ray and MRI examinations of lumbar will be completed to evaluate the imaging manifestations of the responsible and adjacent segments before surgery. Patients with asymptomatic pre-existing canal stenosis factors (cerebrospinal fluid occlusion grade 1) at L3/4 segment will be enrolled. Patients will be randomly divided into two groups according to different strategies. NS Group includes patients who simply receive responsible segments fused (L4-S1). LD Group includes patients who receive responsible segments fused (L4-S1) plus limited decompression at adjacent segment (L3/4). In terms of limited decompression at the adjacent segment, partial laminotomy, flavectomy, and bilateral medial facetectomies up to the pedicle will be performed. Complete laminectomy and destroy of posterior ligament complex will be avoided.

The patient's age, gender, preoperative body mass index (BMI), American Society of Anesthesiologists classification of anesthesia (ASA grade) will be recorded during the hospital stay. Surgical data including operation time, blood loss, perioperative complications (including cerebrospinal fluid leakage, wound infection, postoperative neurological dysfunction, and perioperative secondary surgery, cardiopulmonary complication, cerebral infarction/hemorrhage, etc.), and length of hospital stay are also recorded. Preoperative clinical function questionnaires, including visual analog scale (VAS) of low back, VAS of the legs, and Oswestry Disability Index (ODI) scores for patients were completed on admission for surgery without any assistance. All the patients enrolled will finished the follow-up from date of surgery at 1,2, 5 and 10 years. The clinical outcomes and ASP will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* A clear diagnosis of lumbar spinal stenosis, and surgical level of L4-S1 (The levels to be operated on were decided by matching the clinical symptomatology with the radiological findings of the spinal levels that needed decompression);
* Patients have asymptomatic pre-existing spinal canal stenosis (cerebrospinal fluid occlusion grade=1) at adjacent segment.
* Failed at least eight weeks conservative treatment;

Exclusion Criteria:

* Unstable factors (slip, rotation, lateral bending, etc.) in adjacent segment L3/4;
* Preoperative sagittal and coronal imbalance of the spine;
* Lumbar infection and/or tumor diseases;
* A previous history of lumbar fusion surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2032-08-01 (Estimated)

PRIMARY OUTCOMES:
Adjacent segment degeneration | 12 months after surgery
  ASDeg is defined as follows according to manifestations on X-rays and MRI changing from baseline : (1) Progression ≥1 grade in SCS or L3/4 disc degeneration; (2)Alteration of L3/4 disc herniation, Hiz and vacuum sign; (3) Progression of ≥ 3 mm in vertebral slippage, a change of ≥ 10° in the intervertebral angle on flexion and extension lateral radiograph, or scoliosis deformity on coronal plane.
Adjacent segment degeneration | 24 months after surgery
  ASDeg is defined as follows according to manifestations on X-rays and MRI changing from baseline : (1) Progression ≥1 grade in SCS or L3/4 disc degeneration; (2)Alteration of L3/4 disc herniation, Hiz and vacuum sign; (3) Progression of ≥ 3 mm in vertebral slippage, a change of ≥ 10° in the intervertebral angle on flexion and extension lateral radiograph, or scoliosis deformity on coronal plane.
Adjacent segment degeneration | 60 months after surgery
  ASDeg is defined as follows according to manifestations on X-rays and MRI changing from baseline : (1) Progression ≥1 grade in SCS or L3/4 disc degeneration; (2)Alteration of L3/4 disc herniation, Hiz and vacuum sign; (3) Progression of ≥ 3 mm in vertebral slippage, a change of ≥ 10° in the intervertebral angle on flexion and extension lateral radiograph, or scoliosis deformity on coronal plane.
Adjacent segment degeneration | 120 months after surgery
  ASDeg is defined as follows according to manifestations on X-rays and MRI changing from baseline : (1) Progression ≥1 grade in SCS or L3/4 disc degeneration; (2)Alteration of L3/4 disc herniation, Hiz and vacuum sign; (3) Progression of ≥ 3 mm in vertebral slippage, a change of ≥ 10° in the intervertebral angle on flexion and extension lateral radiograph, or scoliosis deformity on coronal plane.
Adjacent segment disease | The entire study process, up to 120 months after surgery.
  ASDis is defined as clinical and radiographic evidence of degenerative spinal disease (disc degeneration, stenosis, or spondylolisthesis) on the level adjacent to the index fusion.

SECONDARY OUTCOMES:
Disability | 12 months after surgery; 24 months after surgery; 60 months after surgery; 120 months after surgery.
  The Oswestry Disability Index (ODI) (0-100) is used to assess disability.
Back pain | 12 months after surgery; 24 months after surgery; 60 months after surgery; 120 months after surgery.
  The Visual Analog Scale (0-10) is used to evaluate back pain.
Leg pain | 12 months after surgery; 24 months after surgery; 60 months after surgery; 120 months after surgery.
  The Visual Analog Scale (0-10) is used to evaluate leg pain.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Shi Li, Dr., Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
We will make the clinical study report available for half a year after the publication of the results of the study.
Supporting Information: CSR
Time Frame: The IPD will become available for half a year after the publication of the results of the study.
Access Criteria: The IPD is available to the readers of the journal in which our research is published. The corresponding author of the published papers will review the requests.

REFERENCES:
- [Result] Lawrence BD, Wang J, Arnold PM, Hermsmeyer J, Norvell DC, Brodke DS. Predicting the risk of adjacent segment pathology after lumbar fusion: a systematic review. Spine (Phila Pa 1976). 2012 Oct 15;37(22 Suppl):S123-32. doi: 10.1097/BRS.0b013e31826d60d8. PMID 22885827
- [Result] Zhong ZM, Deviren V, Tay B, Burch S, Berven SH. Adjacent segment disease after instrumented fusion for adult lumbar spondylolisthesis: Incidence and risk factors. Clin Neurol Neurosurg. 2017 May;156:29-34. doi: 10.1016/j.clineuro.2017.02.020. Epub 2017 Feb 27. PMID 28288396
- [Result] Alentado VJ, Lubelski D, Healy AT, Orr RD, Steinmetz MP, Benzel EC, Mroz TE. Predisposing Characteristics of Adjacent Segment Disease After Lumbar Fusion. Spine (Phila Pa 1976). 2016 Jul 15;41(14):1167-1172. doi: 10.1097/BRS.0000000000001493. PMID 26863261
- [Result] Hikata T, Kamata M, Furukawa M. Risk factors for adjacent segment disease after posterior lumbar interbody fusion and efficacy of simultaneous decompression surgery for symptomatic adjacent segment disease. J Spinal Disord Tech. 2014 Apr;27(2):70-5. doi: 10.1097/BSD.0b013e31824e5292. PMID 22460400
- [Result] Matsumoto T, Okuda S, Nagamoto Y, Sugiura T, Takahashi Y, Iwasaki M. Effects of Concomitant Decompression Adjacent to a Posterior Lumbar Interbody Fusion Segment on Clinical and Radiologic Outcomes: Comparative Analysis 5 Years After Surgery. Global Spine J. 2019 Aug;9(5):505-511. doi: 10.1177/2192568218803324. Epub 2018 Oct 8. PMID 31431873
- [Result] Lee GY, Lee JW, Choi HS, Oh KJ, Kang HS. A new grading system of lumbar central canal stenosis on MRI: an easy and reliable method. Skeletal Radiol. 2011 Aug;40(8):1033-9. doi: 10.1007/s00256-011-1102-x. Epub 2011 Feb 1. PMID 21286714
- [Result] Nakashima H, Kawakami N, Tsuji T, Ohara T, Suzuki Y, Saito T, Nohara A, Tauchi R, Ohta K, Hamajima N, Imagama S. Adjacent Segment Disease After Posterior Lumbar Interbody Fusion: Based on Cases With a Minimum of 10 Years of Follow-up. Spine (Phila Pa 1976). 2015 Jul 15;40(14):E831-41. doi: 10.1097/BRS.0000000000000917. PMID 25839385